CLINICAL TRIAL: NCT05251324
Title: The Cardiovascular Impact of Hot Flushes
Status: Recruiting | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: STUDY00013742
Record Dates: First submitted 2022-01-04; First posted 2022-02-22 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Hot Flashes; Menopause
Keywords: Menopause
MeSH Terms: conditions — Hot Flashes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Participants With Hot Flushes (at least 3 per day): At Visit 1, participants will complete informed consent, questionnaires regarding medical history, physical activity levels, stress and anxiety, menopause symptoms and a hot flush behavior scale. Visit one will be completed remotely using a HIPAA-compliant online platform or over the phone.
  At Visit 2, baseline measurements will be recorded for two hours and spontaneous hot flushes will be detected. Participants will then have a temperature-controlled, water-circulating heating pad at a consistent temperature of 107˚F placed on their torso for 30 min, followed by five min of recovery. This will be followed by a blood draw to measure sex hormones. At either Visit 2 or a separate visit, participants will have a dual energy x-ray absorptiometry scan for a body composition assessment. For participants taking prescribed MHT, a standard protocol for enrollment and they may complete up to six study visits.
  Interventions: Other: Hot Flush Induction
- Participants Without Hot Flushes: At Visit 1, participants will complete informed consent, questionnaires regarding medical history, physical activity levels, stress and anxiety, menopause symptoms and a hot flush behavior scale. Visit one will be completed remotely using a HIPAA-compliant online platform or over the phone.
  At Visit 2, baseline measurements will be recorded for two hours and spontaneous hot flushes will be detected. Participants will then have a temperature-controlled, water-circulating heating pad at a consistent temperature of 107˚F placed on their torso for 30 min, followed by five min of recovery. This will be followed by a blood draw to measure sex hormones. At either Visit 2 or a separate visit, participants will have a dual energy x-ray absorptiometry scan for a body composition assessment. For participants taking prescribed MHT, a standard protocol for enrollment and they may complete up to six study visits.
  Interventions: Other: Hot Flush Induction

INTERVENTIONS:
Other: Hot Flush Induction — A temperature-controlled, water-circulating heating pad at a constant temperature of 107˚F will be placed on the participant's torso, a microwaved heating neck pad will be placed on the participant's neck, and two warm balloons will be placed in the participant's hands for 30 min. Subjective (verbal start and end point to be marked on LabChart software) and objective (skin conductance and skin temperature) measures of hot flushes will be recorded.

SUMMARY:
The overall objective of this study is to examine the physiological responses that occur during a hot flush in postmenopausal women. The following specific aims will be executed to reach the overall objective of this study. Aim 1: To determine if hot flushes can be reliably induced with a temperature-controlled, water- circulating (TCWC) heating pad. Based on previous research, the investigators hypothesize that hot flushes will be inducible with the TCWC in symptomatic women, but not in asymptomatic women. Aim 2: To determine if heat-induced hot flushes in symptomatic women will cause reproducible cardiovascular and respiratory responses. The investigators hypothesize that heat-induced hot flushes produce similar and reproducible cardiovascular and respiratory responses to spontaneous hot flushes. Aim 3: To determine if body fat percentage influences hot flush severity or frequency during spontaneous or induced hot flushes. The investigators hypothesize that women with higher body fat have reduced hot flash severity and frequency.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) increases aggressively after menopause and is the leading cause of mortality in women in the US. Autonomic dysregulation and high blood pressure (BP), often demonstrated in postmenopausal women, are directly linked to CVD. Women who experience vasomotor symptoms (VMS) of menopause, such as night sweats or hot flushes, are at an increased CVD risk. For example, VMS were associated with endothelial dysfunction, elevated blood pressure (BP) and cholesterol, suggesting that VMS may be a marker of adverse vascular changes associated with CVD. Thus, the investigators have designed a pilot study to 1) replicate the hot flush induction protocol and 2) determine if the cardiovascular responses (increased blood pressure and heart rate) during hot flushes are altered. The investigators hypothesize that VMS, and in particular, hot flushes, will cause elevated BP and HR compared with asymptomatic women. These findings will provide important information to physiological responses of VMS in women, which will provide mechanistic insight to the greater cardiovascular risk observed in women who report these symptoms compared with asymptomatic women.

Hot flushes are the most common symptom of climacteric and are reported as feelings of intense warmth along with sweating, flushing and chills. Indeed, it is suggested that 50-80% of women post-menopause will experience hot flushes. Hot flushes usually last for one to five minutes but can last up to an hour. The median duration of symptoms is about four years, but some can last as long as 20 years. Although estrogen withdrawal is necessary to produce a hot flush, it is not sufficient to explain the occurrence of them as some women do not experience them, but all women experience a deficit in estradiol and progesterone during menopause. There are also no relationships between symptoms and plasma, urinary, or vaginal levels of estrogens, nor are there differences in plasma levels between women with and without hot flushes. The putative physiological trigger of hot flashes is core body temperature elevations acting within a reduced thermoneutral zone. This reduction appears to be closely related to increased central nervous levels of norepinephrine (NE), partly through alpha 2 -adrenergic receptors. The involvement of NE in central thermoregulation and the etiology of hot flushes are supported by results from experimental and animal studies that demonstrate increased central nervous system NE levels narrow the width of the thermoneutral zone. During hot flushes, skin temperature increases in digits, face, arms, chest, abdomen, back and legs; sweating often occurs; and heart rate increases. In previous research, measurable sweating occurred in 90% of hot flushes. Sweat rate corresponds closely to skin conductance, the electrical measure of sweating, during hot flushes. Indeed, sternal skin conductance and skin temperature are the gold standard objective measurement of a hot flush.

Body weight and adiposity are increased by estrogen deficiency, thus estradiol may have a protective role against increased body fat in aging women. In addition, fat mass increases as a consequence of aging and menopause in females. However, aromatase, the rate limiting enzyme of androgen to estradiol conversion, is mainly produce in adipocytes (fat cells), where it becomes an important source for estradiol in the postmenopausal period. Thus, the varying levels of estradiol could influence hot flushes in women. Thus, it is important to characterize fat mass in postmenopausal women to determine if body fat percentage influences the severity or frequency of VMS, either spontaneous or induced.

Hot flushes occur spontaneously, which can make it challenging to measure their etiology and physiological responses to them. Because these vasomotor symptoms are strongly connected with CVD, it is important to understand the mechanism by which these symptoms may lead to CVD. Thus, being able to reliably induce a hot flush is key to understanding these mechanisms. Previous research has demonstrated that hot flushes can be induced pharmacologically with yohimbine, an alpha 2 -adrenergic antagonist, and with controlled heating to the torso in symptomatic women, but not asymptomatic women. While measuring physiological responses to hot flushes, the investigators will be able to determine factors that contribute to the greater CVD risk in women who experience VMS.

Importantly, being able to compare the responses of hot flushes to the predictable and known responses to the cold pressor test. The investigators' central hypothesis is that hot flushes can be induced in symptomatic women with a temperature controlled, water heating pad and that BP and HR will be elevated in these women compared with asymptomatic women. If these findings prove to be true, it suggests that women who have vasomotor symptoms may also demonstrate exaggerated responses to stress and this may be occurring frequently in women who experience these debilitating menopausal symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal (may have or may not have hot flushes)
* Have not started hormone therapy and/or will discontinue hormone therapy for the duration of the study

Exclusion Criteria:

* Reported nicotine/tobacco use within the last six months
* Diabetic or asthmatic
* Diagnosed significant carotid stenosis
* History of significant autonomic dysfunction, heart disease, respiratory disease, or severe neurologic condition such as stroke or traumatic brain injury
* Existing metabolic or endocrine abnormalities
* Use of heart/blood pressure medications that are determined to interfere with study outcomes
* Unwilling to discontinue use of OC (or other hormonal contraceptives, including intrauterine devices or contraceptive implants) and/or MHT
* Pregnant or breastfeeding
* Unwilling or unable to refrain from consuming caffeine or alcohol in the 12 hours before visit two or three
* Unwilling or unable to refrain from vigorous exercise (at least 10 minutes in duration) in the 12 hours before visit two or three
* Unwilling or unable to fast in the eight hours before visit two or three
* Body mass index greater than or equal to 35 kg/m^3

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 40-70-year-old postmenopausal women who experience hot flushes and those who do not.
  Women who have not started hormone therapy and/or will discontinue hormone therapy for the duration of the study.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2026-05-26 (Estimated); Study Completion 2026-05-26 (Estimated)

PRIMARY OUTCOMES:
Systolic Blood pressure (mmHg) | 3 hours
  Blood pressure will be measured using a non-invasive blood pressure cuff and measured in units of mmHG and assessed at Visit 2.
Diastolic Blood pressure | 3 hours
  Blood pressure will be measured using a non-invasive blood pressure cuff and measured in units of mmHG and assessed at Visit 2.
Mean arterial Blood pressure | 3 hours
  Blood pressure will be measured using a non-invasive blood pressure cuff and measured in units of mmHG and assessed at Visit 2.
Skin conductance | 3 hours
  Skin conductance is measured using galvanic skin response and is measured in umho. Skin conductance will be assessed at Visit 2.
Skin temperature | 3 hours
  Skin temperature will be measured by a skin thermometer and reported in °C or °F as an objective measure of hot flushes. Skin temperature will be assessed at Visit 2.

SECONDARY OUTCOMES:
Heart rate | 3 hours
  Heart rate will be measured with a three lead electrocardiogram and measured in beats-per minute Heart rate will be assessed at Visit 2.
Respiratory rate | 3 hours
  Respiratory rate will be measured a respiratory belt and reported in breaths per minute. Respiratory rate will be assessed at Visit 2.
Heart rate variability | 3 hours
  Heart rate will be measured with a three lead electrocardiogram and reported in units of Hertz and milliseconds. Heart rate variability will be assessed at Visit 2.
Numerical pain rating scale | 3 hours
  The numerical pain rating scale consists of 1 item with scores ranging from 1-10, where higher scores represent greater pain. The numerical pain rating scale will be assessed at Visit 2.
Blood levels of estradiol (E2) | 3 hours
  Blood levels of estradiol will be reported as ng/dL. Blood levels of estradiol will be assessed at Visit 2.
Blood levels of estrone (E1) | 3 hours
  Blood levels of estrone will be reported as ng/dL. Blood levels of estrone will be assessed at Visit 2.
Blood levels of total estrogens | 3 hours
  Blood levels of total estrogens will be reported as ng/dL. Blood levels of total estrogens will be assessed at Visit 2.
Blood levels of progesterone | 3 hours
  Blood levels of progesterone will be reported as ng/mL. Blood levels of progesterone will be assessed at Visit 2.
Blood levels of testosterone | 3 hours
  Blood levels of testosterone will be reported as ng/dL. Blood levels of testosterone will be assessed at Visit 2.
Blood levels of Follicle Stimulating Hormone (FSH) | 3 hours
  Blood levels of FSH will be reported as IU/L. Blood levels of FSH will be assessed at Visit 2.
Blood levels of Hemoglobin A1C (HbA1c) | 3 hours
  Blood levels of HbA1c will be reported as g/dL. Blood levels of HbA1c will be assessed at Visit 2.
Menopause-Specific Questionnaire of Life (MENQOL) | 60 minutes
  MENQOL is 29 total items asking about Menopause symptoms, first asking a yes or no question of if they experience the symptoms, and if yes, converted to a 1-7 scale, with 1 indicating less bothersome and 7 indicating more bothersome symptoms. Total scores range from 29-232, where higher scores indicate more bothersome menopause symptoms. MENQOL will be assessed at Visit 1.
State Trait Anxiety Index (STAI) | 60 minutes
  The STAI consists of 20 questions ranging from 1 to 4 (4 representing the most anxiety) with a total score between 20 to 80, where higher summed scores indicate greater anxiety. STAI will be assessed at Visit 1.
Dual x-ray absorptiometry (DXA) of fat mass | 30 minutes during separate visit
  Fat mass measured via DXA will be reported as g/kg. DXA of fat mass will be assessed at Visit 2.
Vitamin D Intake | 15 minutes during separate visit
  Vitamin D intake with be reported as a binary 'yes' or 'no' determined by participant report of Vitamin D supplementation. Vitamin D intake will be assessed at Visit 2.

CONTACTS AND LOCATIONS:
Overall Officials: Manda Keller-Ross, PhD, DPT, PT, Principal Investigator — University of Minnesota Medical School Department of Rehabilitation Medicine
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No